CLINICAL TRIAL: NCT06953310
Title: Assessing the Effects of a Multisectoral Agricultural Intervention on the Reproductive and Sexual Health of Adolescent Girls and Young Women
Acronym: Vijana Shamba
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01MH138256 (NIH); R01MH138256 (NIH)
Record Dates: First submitted 2025-04-17; First posted 2025-05-01 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Sexually Transmitted Infection (STI); HIV; Food Insecurity; Mental Health
Keywords: multisectoral agriculture intervention; sexual and reproductive health; Kenya; adolescent girls and young women; HIV; food insecurity; Shamba Maisha
MeSH Terms: conditions — Sexually Transmitted Diseases; Psychological Well-Being; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shamba Maisha Intervention (Experimental): The Shamba Maisha Intervention inervention has three key parts:
  1. Farming Equipment and Training: The study provide families with water pumps, seeds, and other farming tools to improve their ability to grow food. Caregivers and girls will also get training on how to use these tools.
  2. School-based Farming: Girls will participate in practical farming activities at school, where they can learn and practice the farming skills. This also benefits the entire school because the crops grown can be used to provide food for students.
  3. Caregiver and Adolescent Relationship Strengthening: Families will take part in special sessions where they will learn how to improve their communication, reduce stress, and talk about important topics like sexual health.
  Interventions: Other: Shamba Maisha
- Control Arm (No Intervention): Control participants and schools randomized to the control condition will have the opportunity to receive the full intervention at the conclusion of data collection.

INTERVENTIONS:
Other: Shamba Maisha — The Shamba Maisha Intervention intervention has three key parts:
  Farming Equipment and Training: The study will provide families with water pumps, seeds, and other farming tools to improve their ability to grow food. Caregivers and girls will also get training on how to use these tools.
  School-based Farming: Girls will participate in practical farming activities at school, where they can learn and practice the farming skills. This also benefits the entire school because the crops grown can be used to provide food for students.
  Caregiver and Adolescent Relationship Strengthening: Families will take part in special sessions where they will learn how to improve their communication, reduce stress, and talk about important topics like sexual health.
  Arms: Shamba Maisha Intervention

SUMMARY:
In Kenya, HIV incidence among adolescent girls and young women (AGYW) ages 15-24 years is 1-2 per 100 person-years and approximately 30% of AGYW have had at least one sexually transmitted infection (STI). Kisumu and Migori counties in Western Kenya have some of the highest HIV/STI incidence in the country. Food insecurity (FI) and poverty are also highly prevalent in Western Kenya. FI and poverty are important drivers of vulnerability to HIV and STIs among AGYW. Poverty alleviation interventions have the potential to reduce STIs and HIV risk among AGYW but, to date, these interventions have reported mixed findings on HIV/STI outcomes, have been primarily targeted at the individual level, and none have focused on agriculture or FI. Therefore, there remains a critical need to develop sustainable, multi-level, economic and FI interventions that improve AGYW STI/HIV prevention outcomes. Our team has successfully developed a household-level agricultural intervention in Western Kenya called Shamba Maisha ("farm life" in Kiswahili; SM) to reduce household FI. In our prior pilot study with AGYW, the investigators found that SM was feasible, acceptable, and associated with less FI and improved mental health. In this proposal, the investigators will build upon our promising SM work by examining the effectiveness and implementation of our SM intervention, including provision of a water pump and agricultural implements for use at home, training in agriculture delivered at school-based demonstration farms, and adolescent-caregiver relationship strengthening training. The investigators plan to conduct this school- and home-based cluster randomized trial with 800 AGYW and their primary caregivers recruited from schools in Kisumu and Migori counties. The investigators will randomize 20 schools in Kisumu and Migori in a 1:1 ratio to intervention or control conditions and follow AGYW-caregiver dyads for 18 months with surveys and STI/pregnancy testing to assess intervention impacts. The study has the following aims: Aim 1. Determine the impact of SM on adolescent HIV prevention and sexual and reproductive health outcomes (primary outcome is gonorrhea and/or chlamydia incidence). Aim 2. Assess the effect of SM on intermediate outcomes theorized from our published conceptual framework to be on the causal pathway, including household food security and wealth, and adolescent and caregiver factors including mental health and aspects of the caregiver-AGYW relationship dyad (e.g., communication). Aim 3. Identify critical implementation facilitators and barriers influencing SM effectiveness and delivery and conduct a programmatic cost assessment. The investigators will also evaluate the extent to which SM can have "spillover" nutritional benefits for a larger population of adolescents who had access to demonstration farms at intervention schools but did not receive other aspects of the intervention. The ultimate goal is to provide an innovative household-level intervention to halt the cycle of FI, and poor HIV-related outcomes among vulnerable populations including AGYW, consistent with the "Ending the HIV Epidemic".

ELIGIBILITY:
Inclusion Criteria:

Adolescent Girls and Young women (AGYW):

* AGYW assigned female at birth
* Between 15-19 years of age at enrollment
* Attending the selected schools with at least 18 months remaining of schooling
* STI-uninfected and not pregnant at baseline
* Has an adult caregiver willing to participate
* Demonstrates moderate to severe FI based on the Household Food Insecurity Access Scale (HFIAS), and/or malnutrition (BMI less than two standard deviations below the mean for age-specific BMI

Caregiver:

* At least 18 years old.
* At least 1 AGYW aged 15-19 years old attending the selected schools
* household has access to farming land
* household has available surface water in the form of lakes, rivers, ponds, or shallow wells (home is 200m from permanent water source)

Exclusion Criteria:

* AGYW or adult caregivers who have inadequate cognitive and/or hearing capacity to complete planned study procedures
* AGYW or adult caregivers who do not speak Dholuo, Kiswahili, or English
* Married AGYW and those who serve as heads of households
* AGYW who are pregnant at screening

Adolescent girls who test positive for gonorrhea or chlamydia at screening will be invited to re-screen at least 14 days after receiving treatment and will be eligible to enroll if they have a confirmatory negative STI test.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
STI Incidence (gonorrhea and/or chlamydia incidence) | 0, 6, 12, and 18 months
  Biologic samples
Food insecurity - Household Food Insecurity Access Scale (HFIAS). | 0, 6, 12, 18 months
  Household Food Insecurity Access Scale (HFIAS). Scores ranges from 0-27, with higher scores indicating higher food insecurity.
Depression among adolescents - Patient Health Questionnaire - 9 (PHQ-9) | 0, 6, 12, and 18 months
  Patient Health Questionnaire - 9 (PHQ-9) among adolescents. Scores range from 0 - 27, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Body Mass Index (BMI) among adolescents | 0, 6, 12, 18 months
  Body Mass Index (BMI) among adolescents
Depression among caregivers - Patient Health Questionnaire - 9 (PHQ-9) | 0, 6, 12, 18 months
  Patient Health Questionnaire - 9 (PHQ-9) among caregivers. Scores range from 0 - 27, with higher scores indicating more severe depression.
Anxiety among adolescents - General Anxiety Disorder-7 (GAD-7) | 0, 6, 12, 18 months
  General Anxiety Disorder-7 (GAD-7) among adolescents. Scores range from 0 - 21, with higher scores indicating more severe anxiety.
Pregnancy rate among adolescents | 0, 6, 12, 18 months
  Pregnancy rate among adolescents
Percent of sexually active adolescents who self-report condom use | 0, 6, 12, 18 months
  Percent of sexually active adolescents who self-report condom use
WHO Domestic Violence Module - Intimate Partner Violence among adolescents | 0, 6, 12, 18 months
  WHO Domestic Violence Module. Includes physical violence, sexual violence, and emotional abuse. Scores range from 0 to 52 with higher scores indicating more violence.
Parent-child communication | 0, 6, 12, 18 months
  Parent-child communication: Families Matter! Program Tool
Empowerment (Self-esteem) among adolescents - Rosenberg Self-Esteem Scale (RSES) | 0, 6, 12, 18 months
  The Rosenberg Self-Esteem Scale (RSES). The scale ranges from 0-30, with higher scores indicating higher self-esteem.
Educational attainment among adolescents | 0, 6, 12, 18 months
  Self-Reported School attendance

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Weiser, MD, MPH, Principal Investigator — University of California, San Francisco; Jennifer Velloza, PhD, MPH, Principal Investigator — University of California, San Francisco; Maricianah Onono, MBChB, MS, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute (KEMRI), Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual participant data (IPD) in The National Institute of Mental Health Data Archive (NDA) and the SAP and source code will be available in a GitHub repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available by May 2029
Access Criteria: The investigators will share IPD and supporting information upon reasonable request from the scientific community. Source code will be available on a GitHub repository along with a codebook and description of the SAP. A link to the repository will be available after requests are reviewed and approved by the investigator team.

REFERENCES:
- [Background] Cohen CR, Weke E, Frongillo EA, Sheira LA, Burger R, Mocello AR, Wekesa P, Fisher M, Scow K, Thirumurthy H, Dworkin SL, Shade SB, Butler LM, Bukusi EA, Weiser SD. Effect of a Multisectoral Agricultural Intervention on HIV Health Outcomes Among Adults in Kenya: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2246158. doi: 10.1001/jamanetworkopen.2022.46158. PMID 36508217
- [Background] Onono MA, Sheira L, Frongilio EA, Odhiambo G, Wekesa P, Conroy A, Bukusi EA, Cohen CR, Weiser SD. Effect of improving food security on parenting practices and caregiver-adolescent relationships: qualitative findings of an income-generating agricultural intervention in rural Kenya. BJPsych Open. 2024 Dec 26;11(1):e10. doi: 10.1192/bjo.2024.802. PMID 39721953
- [Background] Onono MA, Frongillo EA, Sheira LA, Odhiambo G, Wekesa P, Conroy AA, Cohen CR, Bukusi EA, Weiser SD. Links between Household-Level Income-Generating Agricultural Intervention and the Psychological Well-Being of Adolescent Girls in Human Immunodeficiency Virus-Affected Households in Southwestern Kenya: A Qualitative Inquiry. J Nutr. 2023 Dec;153(12):3595-3603. doi: 10.1016/j.tjnut.2023.10.008. Epub 2023 Oct 18. PMID 37863268
- [Background] Onono MA, Odhiambo G, Sheira L, Conroy A, Neilands TB, Bukusi EA, Weiser SD. The role of food security in increasing adolescent girls' agency towards sexual risk taking: qualitative findings from an income generating agricultural intervention in southwestern Kenya. BMC Public Health. 2021 Nov 6;21(1):2028. doi: 10.1186/s12889-021-12051-6. PMID 34742285
- See also: Related Info — https://shambamaisha.ucsf.edu/